CLINICAL TRIAL: NCT03958097
Title: A Pilot Study of NK Cell Combined With PD-1 Antibody as Second Line Therapy for Advanced Driver Mutation Negative Non-small Cell Lung Cancer
Brief Title: Natural Killer(NK) Cell Combined With Programmed Death-1(PD-1) Antibody as Second Line Therapy for Advanced Driver Mutation Negative Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19K047-001
Record Dates: First submitted 2019-05-20; First posted 2019-05-21 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: sintilimab plus NK cell
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NK cell combined with PD-L1 antibody (Experimental): Autologous peripheral blood mononuclear cells (PBMCs) are collected by apheresis on D0, then induced into NK cells and infused into the patients 14 days later (D14) as the initial transfusion. There are 3 consecutive transfusion days (D14-D16), total NK cells infused at least 3×10^9 .
  200mg PD-L1 antibody(Sintilimab Injection) will be given on D14, 1 hour after NK cells infusion.
  NK cells and PD-L1 antibody will be infused every 21 days until disease progression or unacceptable adverse events.
  Interventions: Combination Product: NK cell and PD-1 antibody

INTERVENTIONS:
Combination Product: NK cell and PD-1 antibody — Each patient enrolled the study will received both NK cell and PD-1 antibody.

SUMMARY:
PD-1 antibody has been approved as second line therapy for driven mutation negative non-small cell lung cancer, but overall response rate is only between 15-20%. Basic study found NK cell can enhance anti-tumor ability of PD-L1 antibody. This study evaluates the efficacy and safety of NK cell combined with PD-1 antibody for advanced driven mutation negative non-small cell lung cancer (NSCLC) as second-line therapy.

DETAILED DESCRIPTION:
The incidence of non-small cell lung cancer is high, and most patients are in advanced stage at the time of diagnosis, and the overall prognosis is poor. Currently, patients with advanced non-small cell lung cancer are treated individually according to the molecular and histological features of the tumor. For patients with negative driver mutation in epidermal growth factor receptor(EGFR), anaplastic lymphoma kinase(ALK),ROS proto-oncogene1(ROS1), v-raf murine sarcoma viral oncogene homolog B1(BRAF) and other driving genes, platinum-based dual chemotherapy combined with PD-1/PD-L1 monoclonal antibody is recommended for first-line treatment. In patients who have not used PD-1/PD-L1 antibody in first-line therapy, the second-line treatment regimen is the first choice for the recommended single-agent PD-1/PD-L1 antibody. However, the current efficacy of PD-1/PD-L1 antibody for second-line treatment of advanced non-small cell lung cancer is limited, only between 15-20%. NK cells secrete interferon(IFN) to promote the expression of PD-L1 in tumor cells and enhance the role of PD-1 inhibitors. At the same time, PD-1 antibodies can bind to NK cell surface PD-1, prevent NK cell depletion, and enhance NK cell anti-tumor. Therefore, the application of NK cells combined with PD-1 antibody in the treatment of patients with advanced non-small cell lung cancer may achieve better results.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age ≥ 18 years old.
* (2) Locally advanced (IIIB/IIIC phase) or metastatic NSCLC (squamous or non-squamous) confirmed by histological examination.
* (3) Disease progression occurred after platinum-based chemotherapy in the previous line, and measurable lesions existed according to RECIST v1.1.
* (4) Patients must be able to provide fresh or archived tumor tissue and pathology reports. Non-squamous NSCLC must be able to provide a report that is confirmed to be wild-type EGFR by tissue-based assays.
* (5) Eastern Cooperative Oncology Group(ECOG) performance status(PS) ≤ 1.
* (6) The vital organs are fully functional, and the following results are obtained for each laboratory indicator (accepting the results of the examinations made within ≤ 28 days before randomization):

  * Cardiac ultrasound indicates a cardiac ejection fraction ≥ 50%; blood oxygen saturation ≥ 90%;
  * Absolute neutral cell count (ANC) ≥ 1.5 x 109/L, platelet count ≥ 100 x 109/L, hemoglobin ≥ 90g/dL;
  * Creatinine (Cr) ≤ 2.5 times normal range;
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 times normal range, total bilirubin (TBIL) ≤ 1.5 times normal range.
* (7) No contraindications for apheresis and cell separation.
* (8) Male or female with fertility needs to agree to take effective contraceptive measures during the study period and at least 120 days after the end of medication.
* (9) A written informed consent can be provided and the research requirements are understood and followed.

Exclusion Criteria:

* (1) Previously received immunological checkpoint inhibitors targeting PD-1, PD-L1 or C ytotoxic T - L ymphocyte A ntigen 4(CTLA-4) and other immunotherapies (including but not limited to interferon or IL-2, chimeric antigen receptor T Cells, vaccines, etc.).
* (2) NSCLC with EGFR gene mutation or ALK gene translocation.
* (3) The toxicity caused by previous anticancer treatment has not recovered to baseline level or returned to stability (except for hair loss, rash, pigmentation or specific laboratory abnormalities).
* (4) A history of severe allergic reactions to other monoclonal antibodies.
* (5) History of interstitial pneumonia, non-infectious pneumonia or uncontrolled systemic diseases, including diabetes, hypertension, and pulmonary fibrosis.
* (6) Clinically severe pericardial effusion.
* (7) Pleural effusion or ascites that is clinically uncontrolled and requires thoracentesis or abdominal puncture drainage within 2 weeks prior to randomization.
* (8) Active pia mater disease or unstable brain metastasis.
* (9) Major surgery, open biopsy or severe traumatic injury was performed ≤ 28 days prior to randomization, or major surgical procedures were expected during the study.
* (10) Other malignant tumors other than NSCLC (except for surgically resected non-melanoma skin cancer, fully treated cervical carcinoma in situ, cured local prostate cancer, fully treated low-grade bladder cancer, Curatively treated breast ductal carcinoma in situ, or a malignant tumor diagnosed 2 years ago, but there is currently no evidence of disease in the absence of treatment ≤ 2 years prior to randomization).
* (11) Severe chronic or active infections requiring systemic antibacterial, antifungal or antiviral treatment, including HIV, hepatitis B virus(HBV), hepatitis C virus(HCV) infection.
* (12) Active autoimmune disease or a history of autoimmune disease but may recur.
* (13) Subjects who require systemic treatment with corticosteroids or other immunosuppressive agents within 14 days prior to randomization.
* (14) Those who have undergone organ transplantation or hematopoietic stem cell transplantation.
* (15) Any live vaccine against infectious diseases (eg, influenza, chickenpox, etc.) was used within 28 days prior to randomization.
* (16) Meet any of the following cardiovascular disease criteria:

  * Evidence of acute or positive myocardial ischemia
  * There are currently symptomatic pulmonary embolisms
  * Acute myocardial infarction occurred within ≤6 months before randomization.
  * Has reached the New York Heart Association grading standard (see Appendix 5) 3 or 4 before randomization ≤ 6 months Grade of heart failure.
  * A ≥2 grade ventricular arrhythmia occurred within ≤6 months before randomization.
  * A cerebrovascular accident (CVA) or transient ischemic attack (TIA) occurred within ≤6 months before randomization.
* (17) Pregnant and lactating women.
* (18) If the patient is unable to follow the study procedures, limitations, and requirements, the investigator believes that the patient is not allowed to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-05-17 (Actual); Primary Completion 2020-10-21 (Actual); Study Completion 2021-10-21 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival(PFS) | 12 months
  From the random date until the date when the objective disease progression (evaluated by the investigator according to RECIST 1.1) or for any reason (whichever occurs first) is confirmed, based on the intent to treat(ITT) set.

SECONDARY OUTCOMES:
Overall Response Rate(ORR) | 12 months
  The proportion of patients with complete response(CR) or partial response(PR) (evaluated by the investigator according to RECIST 1.1), based on the ITT set.
Overall Survival(OS) | 12 months
  The time from the random date to the date of death for any reason, based on the ITT population.
Duration of Response(DoR) | 12 months
  The time from the first confirmed objective remission to recurrence (evaluated by the investigator according to RECIST 1.1) or for any reason, whichever occurs first.

OTHER OUTCOMES:
Disease Control Rate(DCR) | 12 months
  The proportion of patients with the best overall response to CR, PR, or disease stabilization (SD) (according to RECIST V1.1 evaluation).
Clinical Benefit Rate(CBR) | 12 months
  The proportion of patients who have achieved CR, PR, or SD for > 24 weeks (according to RECIST 1.1).
Prognostic biomarkers1 | 12 months
  Level of PD-L1 expression on tumor.
Prognostic biomarkers2 | 12 months
  Tumor mutation burden(TMB) number of tumor tissue.
Prognostic biomarkers3 | 12 months
  Level of PD-L1 expression on NK cell.
Prognostic biomarkers4 | 12 months
  Concentration of patients' serum IL-8.
Prognostic biomarkers5 | 12 months
  Concentration of patients' serum lactic dehydrogenase(LDH).

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jia L, Chen N, Chen X, Niu C, Liu Z, Ma K, Wang N, Yang L, Zhao Y, Song W, Lu J, Chen C, Cong X, Wang X, Xu Y, Cui G, Liu Z, Chen R, Li W, Cui J. Sintilimab plus autologous NK cells as second-line treatment for advanced non-small-cell lung cancer previous treated with platinum-containing chemotherapy. Front Immunol. 2022 Dec 8;13:1074906. doi: 10.3389/fimmu.2022.1074906. eCollection 2022. PMID 36569881
- [Derived] Jia L, Chen N, Chen X, Niu C, Liu Z, Ma K, Yang L, Zhao Y, Song W, Lu J, Chen C, Cong X, Wang X, Xu Y, Cui G, Liu Z, Chen R, Yin H, Zhang N, Cui J. Updated overall survival data and predictive biomarkers of autologous NK cells plus Sintilimab as second-line treatment for advanced non-small cell lung cancer. Front Immunol. 2025 May 21;16:1595382. doi: 10.3389/fimmu.2025.1595382. eCollection 2025. PMID 40469279